CLINICAL TRIAL: NCT00953498
Title: Influence of Glitazones on the Vasodilatory Effect of HDL Lipoproteins and on Phospholipase A2
Brief Title: Influence of Glitazones on the Vasodilatory Effect of High-density Lipoprotein (HDL) Lipoproteins
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Principal Investigator, Prof. Bruno Vergès, Professor, Centre Hospitalier Universitaire Dijon
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AFSSAPS A70516-50
Record Dates: First submitted 2009-08-05; First posted 2009-08-06 (Estimated); Last update posted 2013-09-02 (Estimated); Status verified 2013-08

CONDITIONS: Type 2 Diabetes
Keywords: diabetes; glitazones; HDL
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Pioglitazone; Rosiglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pioglitazone (Active Comparator): treatment with pioglitazone (dose from 30 mg:day to 45 mg/day)
  Interventions: Drug: pioglitazone
- rosiglitazone (Active Comparator): treatment with rosiglitazone at a dose between 4mg and 8 mg/day
  Interventions: Drug: rosiglitazone

INTERVENTIONS:
Drug: pioglitazone — After randomization, patients will be treated by pioglitazone or rosiglitazone
  Other Names: pioglitazone: ACTOS; rosiglitazone: AVANDIA
  Arms: pioglitazone
Drug: rosiglitazone — treatment with rosiglitazone at a dose between 4mg and 8 mg/day
  Other Names: pioglitazone: ACTOS; rosiglitazone: AVANDIA
  Arms: rosiglitazone

SUMMARY:
HDL from patients with type 2 diabetes show a significant reduction of their endothelium-dependent vasodilatory effect.

The primary objective of the study is to analyze whether treatment with glitazones (pioglitazone and rosiglitazone)may improve the endothelium-dependent vasodilatory effect of HDL lipoproteins in patients with type 2 diabetes.

The secondary objectives are:

* to analyze the effect of glitazone treatment on phospholipase A2
* to look for possible differences between the effects of pioglitazone and those of rosiglitazone
* to analyze the glycemic response to glitazone therapy according to clinical and biological baseline characteristics.

DETAILED DESCRIPTION:
The study will be performed as follows:

At baseline, before initiating glitazone treatment, clinical data will be recorded and blood samples will be obtained for biological measurements (blood glucose, HbA1c, total cholesterol, triglycerides, LDL-cholesterol, HDL-cholesterol, liver enzymes), phospholipase A2 measurement and the study of the vasodilatory effect of HDL particles.For this purpose, we will study,using rabbit aorta rings,the ability of HDL to suppress the inhibition of vasodilation that is induced by oxidised LDL.

For all the patients included into the study, a treatment by pioglitazone (at an initial dose of 30 mg/day) or rosiglitazone (at an initial dose of 4 mg/day) will be given by randomization.

A visit will be performed at week 12, in order to titrate the glitazone dose (up to 45 mg/day for pioglitazone, up to 8 mg/day for rosiglitazone)according to HbA1c level and values of self-monitoring blood glucose.

At week 24, the last visit will take place. During this visit, clinical data will be recorded and blood samples will be obtained for biological measurements (blood glucose, HbA1c, total cholesterol, triglycerides, LDL-cholesterol, HDL-cholesterol, liver enzymes), phospholipase A2 measurement and the study of the vasodilatory effect of HDL particles.

ELIGIBILITY:
Inclusion Criteria:

* patients with type 2 diabetes treated by oral antidiabetic agents (except glitazones) and/or insulin
* age> 18 years
* HbA1c > 6.5%

Exclusion Criteria:

* renal failure
* heart failure
* primary hyperlipidemia
* pregnancy
* treatment that may modify lipid metabolism (glucocorticoids, oestrogens, retinoids, HIV antiviral drugs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-10; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Action of glitazone on the endothelium-dependent vasodilatory effects of HDL lipoproteins | 6 months

SECONDARY OUTCOMES:
Effect of glitazone therapy on Phospholipase A2 level | 6 months
Analyze the glycemic response to glitazones according to baseline clinical and biological characteristics | 6 months
Look for possible differences between pioglitazone and rosiglitazone for their effects on HDL lipoproteins and phospholipase A2 | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bruno L Vergès, MD,PhD, Principal Investigator — CHU Dijon
Locations (1):
- Service Endocrinologie-diabétologie, Hôpital du Bocage CHU, Dijon, France

REFERENCES:
- [Background] Persegol L, Verges B, Foissac M, Gambert P, Duvillard L. Inability of HDL from type 2 diabetic patients to counteract the inhibitory effect of oxidised LDL on endothelium-dependent vasorelaxation. Diabetologia. 2006 Jun;49(6):1380-6. doi: 10.1007/s00125-006-0244-1. Epub 2006 Apr 5. PMID 16596357
- [Derived] Verges B, Radu L, Baillot-Rudoni S, Brindisi MC, Poussier A, Bouillet B, Petit JM, Duvillard L. Low HDL-cholesterol: a strong predictor of glycemic response to glitazone treatment in patients with type 2 diabetes. Diabetes Res Clin Pract. 2011 Jul;93(1):e44-8. doi: 10.1016/j.diabres.2011.04.005. Epub 2011 May 6. PMID 21529978